CLINICAL TRIAL: NCT07183306
Title: A Clinical Study to Evaluate Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of HT-101 Injection and/or HT-102 Injection in Patients With Chronic Hepatitis B Virus Infection
Brief Title: A Clinical Study of HT-101 and/or HT-102 in Patients With Chronic Hepatitis B Virus Infection
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Suzhou HepaThera Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HT-101&HT-102-101
Record Dates: First submitted 2025-09-05; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Experimental: Cohort A (HT-101) (Experimental): Participants will receive received HT-101 injection, administered once every 4 weeks (Q4W), at least for 24 weeks
  Interventions: Drug: HT-101
- Experimental: Cohort AA (HT-101) (Experimental): Participants will receive received HT-101 injection, administered once every 4 weeks (Q4W), at least for 24 weeks
  Interventions: Drug: HT-101
- Experimental: Cohort B （HT-102；HT-101） (Experimental): Participants will receive HT-102 injection, administered Q4W for 24 weeks and sequential dosed with HT-101 for another 24 weeks
  Interventions: Drug: HT-101; Drug: HT-102
- Experimental: Cohort C (HT-101 + HT-102) (Experimental): Participants will receive HT-101 injection combined with HT-102 injection, administered once every 4 weeks for 24weeks
  Interventions: Drug: HT-101; Drug: HT-102
- Experimental: Cohort D (HT-101 + HT-102) (Experimental): Participants will receive HT-101 injection combined with HT-102 injection, administered once every 4 weeks for 24weeks
  Interventions: Drug: HT-101; Drug: HT-102
- Experimental: Cohort E (HT-101 + HT-102) (Experimental): Participants will receive HT-101 injection combined with HT-102 injection, administered once every 4 weeks for 24weeks
  Interventions: Drug: HT-101; Drug: HT-102

INTERVENTIONS:
Drug: HT-101 — HT-101 given by subcutaneous injection.
Drug: HT-102 — HT-102 given by subcutaneous injection.
  Arms: Experimental: Cohort B （HT-102；HT-101）; Experimental: Cohort C (HT-101 + HT-102); Experimental: Cohort D (HT-101 + HT-102); Experimental: Cohort E (HT-101 + HT-102)

SUMMARY:
This study is A multicenter, open-label, partial multiple-ascending doses phase1b/2 in which participants with chronic hepatitis B virus (HBV) infection will receive HT-101 and/or HT-102 and be assessed for safety, tolerability, Pharmacokinetics, and Pharmacodynamics. Approximately 86 patients with chronic hepatitis B infection were planned to be recruited. Among them, Group A and Group AA received HT-101 injection, administered once every 4 weeks (Q4W), at least for 24 weeks. Group B received HT-102 injection, administered Q4W for 24 weeks and sequential dosed with HT-101 for another 24 weeks. Groups C, D, and E received HT-101 injection combined with HT-102 injection, administered once every 4 weeks for 24weeks. During the study period, all subjects received nucleoside (acid) analogues (NAs) treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects were eligible for inclusion into the study if they met each of the following criteria:

Patient with CHB

Male subjects weighed ≥ 50.0 kg, female subjects weighed ≥ 45.0 kg, with a body mass index (BMI) between 19.0 and 28.0 kg/m^2 (inclusive); Chronic HBV infection for >/= 6 months; The quantitation level of HBsAg was > 100 IU/mL and <3000 IU/mL; The quantitation level of HBV DNA <LLOQ;

· On Nas therapy for >/= 6 months at the time of screening

Subjects promised to use effective contraception for at least 1 month before screening, and have no fertility, donate sperm or eggs and voluntarily take highly effective physical contraception (including partners) during the trial and within 3 months after the end of the trial;

Exclusion Criteria:

* Subjects were excluded from the study if one or more of the following criteria were applicable

Participants with history of drug allergy or specific allergy; Participants who had psychiatric conditions or diseases in cardiovascular, respiratory, endocrine, kidney, liver, digestive tract, skin, immune, blood, nerve and other systems; Participants with history of active pathological bleeding, or bleeding tendency; Participants with abnormal results of physical examination, vital sign examination, ECG examination, laboratory test in the screening period which were judged as clinically significant by clinicians; Participants with significant liver fibrosis or cirrhosis; Participants with symptoms or a history of hepatic decompensation; Participants with a history or suspected risk of liver cancer;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2024-12-30 (Actual); Primary Completion 2026-08-24 (Estimated); Study Completion 2027-05-03 (Estimated)

PRIMARY OUTCOMES:
Clinically significant abnormalities | From enrollment to the end of treatment at up to 60 weeks
  Number of subjects with clinically significant abnormalities in vital signs, electrocardiogram (ECG), and laboratory parameters graded by CTCAE v5.0.
Incidence of adverse events (AEs) and serious adverse events (SAEs) | From enrollment to the end of treatment at up to 60 weeks
  Number of subjects with adverse events (AEs) and serious adverse events (SAEs) assessed by the Common Terminology Criteria for Adverse Events (CTCAE) v5.0.

SECONDARY OUTCOMES:
Maximum Plasma Concentration (Cmax) | HT-101: From predose 1 hour to postdose 24 hours HT-102：UP to 36 weeks
  Cmax of HT-101 and its metabolite in plasma. First administration: Predose 1 hour; Postdose 0.5 hours, 2 hours, 4 hours, 6 hours, 8 hours, 12 hours, 24 hours.
  Changes in the concentration of and HT-102 in serum, From Day1 until 36 weeks
Time to Reach Maximum Plasma Concentration (Tmax) | HT-101：From predose 1 hour to postdose 24 hours. HT-102：UP to 36 weeks
  Tmax of HT-101 and its metabolite in plasma. First administration: Predose 1 hour; Postdose 0.5 hours, 2 hours, 4 hours, 6 hours, 8 hours, 12 hours, 24 hours.
  Changes in the concentration of and HT-102 in serum, From Day1 until 36 weeks
Area Under the Plasma Concentration Versus Time Curve (AUC) | HT-101：From predose 1 hour to postdose 24 hours. HT-102：UP to 36 weeks
  AUC of HT-101 and its metabolite from time 0 to last measurable time. First administration: Predose 1 hour; Postdose 0.5 hours, 2 hours, 4 hours, 6 hours, 8 hours, 12 hours, 24 hours.
  Changes in the concentration of and HT-102 in serum, From Day1 until 36 weeks
Apparent Terminal Elimination Half-life (T1/2) | HT-101：From predose 1 hour to postdose 24 hours. HT-102：UP to 36 weeks
  T1/2 of HT-101 in plasma. First administration: Predose 1 hour; Postdose 0.5 hours, 2 hours, 4 hours, 6 hours, 8 hours, 12 hours, 24 hours.
  Changes in the concentration of and HT-102 in serum, From Day1 until 36 weeks
Apparent Plasma Clearance (CL/F) | HT-101：From predose 1 hour to postdose 24 hours. HT-102：UP to 36 weeks
  CL/F of HT-101 in plasma. First administration: Predose 1 hour; Postdose 0.5 hours, 2 hours, 4 hours, 6 hours, 8 hours, 12 hours, 24 hours.
  Changes in the concentration of and HT-102 in serum, From Day1 until 36 weeks
Apparent volume of distribution（Vd/F） | HT-101：From predose 1 hour to postdose 24 hours. HT-102：UP to 36 weeks
  Vd/F of HT-101. First administration: Predose 1 hour; Postdose 0.5 hours, 2 hours, 4 hours, 6 hours, 8 hours, 12 hours, 24 hours.
  Changes in the concentration of and HT-102 in serum, From Day1 until 36 weeks
Maximum Change of Serum HBsAg From Baseline | Up to 48 weeks
  Maximum change of serum HBsAg from Day 1 until 48 weeks post last dose (negative values mean reductions from baseline, positive values mean increased from baseline)
Maximum Change of Serum HBV DNA From Baseline | Up to 48 weeks
  Maximum change of serum HBV DNA from Day 1 until 48 weeks (negative values mean reductions from baseline, positive values mean increased from baseline).
Titers of Anti-drug Antibody (ADA) to HT-102 | UP to 36 weeks
  ADA analysis for predose 36weeks

CONTACTS AND LOCATIONS:
Locations (7):
- China (7):
  - Beijing Ditan Hospital Capital Medical University, Beijing, Beijing Municipality
  - Xiamen Hospital of Traditional Chinese Medicine, Xiamen, Fujian
  - Guangzhou Eighth People's Hospital, Guangzhou Medical University, Guangzhou, Guangdong
  - Nanfang Hospital, Guangzhou, Guangdong
  - Qingyuan People's Hospital, Qingyuan, Guangdong
  - Shanghai Public Health Clinical Center, Shanghai, Shanghai Municipality
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan